CLINICAL TRIAL: NCT00271739
Title: Informatics for Diabetes Education and Telemedicine (IDEATel)
Brief Title: Randomized Trial of Telemedicine for Diabetes Care
Acronym: IDEATel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Steven J. Shea, Hamilton Southworth Professor of Medicine and Professor of Epidemiology (in Biomedical Informatics); Senior Vice Dean , College of Physicians and Surgeons, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAA5372; CMS 95-C-90998 (Other: protocol)
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus
Keywords: Telemedicine; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemedicine case management (Experimental): Telemedicine visits conducted by a registered nurse (RN) with remote monitoring of blood pressure (BP) and blood glucose through the use of a telemedicine home unit (HTU).
  Interventions: Device: Telemedicine Unit (HTU)
- Usual care (Active Comparator): usual care by primary care provider
  Interventions: Other: usual care

INTERVENTIONS:
Device: Telemedicine Unit (HTU) — This study involves the deployment of a home telemedicine unit (HTU). The HTU provides 3 critical functions for patients: videoconferencing, access to information resources and e-mail through a web-enabled workstation, and medical data acquisition through an electronic device interface. The HTUs also included a glucometer and a blood pressure cuff interfaced directly with the HTU.
  Other Names: HTU
  Arms: Telemedicine case management
Other: usual care — usual diabetes care, as provided by primary care providers
  Arms: Usual care

SUMMARY:
The IDEATel study is a multicenter randomized controlled trial to evaluate the efficacy, acceptability, and cost-effectiveness of telemedicine case management to provide diabetes care to elderly Medicare beneficiaries residing in medically underserved areas of New York State.

DETAILED DESCRIPTION:
The project is designed as a randomized controlled trial with approximately 750 subjects receiving a telemedicine intervention and approximately 750 receiving usual care. Eligibility requires having diabetes, being a Medicare beneficiary, and living in a medically underserved area. The project is conducted in New York City, in northern Manhattan (urban component), and in rural upstate New York through a consortion of participating institutions based at the State University of New York (SUNY) Upstate Medical University at Syracuse (rural component). Subjects are randomized to receive telemedicine case management or usual care for diabetes. The intervention utilizes a home telemedicine unit (HTU). The HTU is a specially designed, web-enabled device with a data port connected to a home glucometer and home blood pressure cuff whereby measurements obtained with these devices can be directly uploaded to a computer database. A diabetes nurse case manager interacts regularly with intervention participants through videoconference via the HTU.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or greater
* Being a current Medicare beneficiary (verified by the Centers for Medicare and Medicaid Services)
* Having diabetes mellitus as defined by a physician's diagnosis and being on treatment with diet, an oral hypoglycemic agent, or insulin
* Residence in a federally designated medically underserved area (either of two federal designations, Medically Underserved Area [MUA] or Health Manpower Shortage Area [HPSA]) in New York Sate
* Fluency in either English or Spanish

Exclusion Criteria:

* Moderate or severe cognitive, visual, or physical impairment
* The presence of severe co-morbid disease.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1665 (Actual)
Dates: Start 2000-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shea, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York

REFERENCES:
- [Background] Shea S, Starren J, Weinstock RS, Knudson PE, Teresi J, Holmes D, Palmas W, Field L, Goland R, Tuck C, Hripcsak G, Capps L, Liss D. Columbia University's Informatics for Diabetes Education and Telemedicine (IDEATel) Project: rationale and design. J Am Med Inform Assoc. 2002 Jan-Feb;9(1):49-62. doi: 10.1136/jamia.2002.0090049. PMID 11751803
- [Background] Starren J, Hripcsak G, Sengupta S, Abbruscato CR, Knudson PE, Weinstock RS, Shea S. Columbia University's Informatics for Diabetes Education and Telemedicine (IDEATel) project: technical implementation. J Am Med Inform Assoc. 2002 Jan-Feb;9(1):25-36. doi: 10.1136/jamia.2002.0090025. PMID 11751801
- [Result] Shea S, Weinstock RS, Starren J, Teresi J, Palmas W, Field L, Morin P, Goland R, Izquierdo RE, Wolff LT, Ashraf M, Hilliman C, Silver S, Meyer S, Holmes D, Petkova E, Capps L, Lantigua RA. A randomized trial comparing telemedicine case management with usual care in older, ethnically diverse, medically underserved patients with diabetes mellitus. J Am Med Inform Assoc. 2006 Jan-Feb;13(1):40-51. doi: 10.1197/jamia.M1917. Epub 2005 Oct 12. PMID 16221935
- [Derived] Palta P, Golden SH, Teresi J, Palmas W, Weinstock RS, Shea S, Manly JJ, Luchsinger JA. Mild cognitive dysfunction does not affect diabetes mellitus control in minority elderly adults. J Am Geriatr Soc. 2014 Dec;62(12):2363-8. doi: 10.1111/jgs.13129. Epub 2014 Nov 29. PMID 25439094
- [Derived] Shea S, Kothari D, Teresi JA, Kong J, Eimicke JP, Lantigua RA, Palmas W, Weinstock RS. Social impact analysis of the effects of a telemedicine intervention to improve diabetes outcomes in an ethnically diverse, medically underserved population: findings from the IDEATel Study. Am J Public Health. 2013 Oct;103(10):1888-94. doi: 10.2105/AJPH.2012.300909. Epub 2013 Mar 14. PMID 23488491
- [Derived] Trief PM, Izquierdo R, Eimicke JP, Teresi JA, Goland R, Palmas W, Shea S, Weinstock RS. Adherence to diabetes self care for white, African-American and Hispanic American telemedicine participants: 5 year results from the IDEATel project. Ethn Health. 2013;18(1):83-96. doi: 10.1080/13557858.2012.700915. Epub 2012 Jul 5. PMID 22762449
- [Derived] Remler DK, Teresi JA, Weinstock RS, Ramirez M, Eimicke JP, Silver S, Shea S. Health care utilization and self-care behaviors of Medicare beneficiaries with diabetes: comparison of national and ethnically diverse underserved populations. Popul Health Manag. 2011 Feb;14(1):11-20. doi: 10.1089/pop.2010.0003. Epub 2011 Jan 17. PMID 21241171
- [Derived] Weinstock RS, Brooks G, Palmas W, Morin PC, Teresi JA, Eimicke JP, Silver S, Izquierdo R, Goland R, Shea S. Lessened decline in physical activity and impairment of older adults with diabetes with telemedicine and pedometer use: results from the IDEATel study. Age Ageing. 2011 Jan;40(1):98-105. doi: 10.1093/ageing/afq147. Epub 2010 Nov 16. PMID 21081539
- [Derived] Homenko DR, Morin PC, Eimicke JP, Teresi JA, Weinstock RS. Food insecurity and food choices in rural older adults with diabetes receiving nutrition education via telemedicine. J Nutr Educ Behav. 2010 Nov-Dec;42(6):404-9. doi: 10.1016/j.jneb.2009.08.001. PMID 21070978
- [Derived] West SP, Lagua C, Trief PM, Izquierdo R, Weinstock RS. Goal setting using telemedicine in rural underserved older adults with diabetes: experiences from the informatics for diabetes education and telemedicine project. Telemed J E Health. 2010 May;16(4):405-16. doi: 10.1089/tmj.2009.0136. PMID 20507198
- [Derived] Robinson KS, Morin PC, Shupe JA, Izquierdo R, Ploutz-Snyder R, Meyer S, Teresi JA, Starren J, Shea S, Weinstock RS. Use of three computer training methods in elderly underserved rural patients enrolled in a diabetes telemedicine program. Comput Inform Nurs. 2010 May-Jun;28(3):172-7. doi: 10.1097/NCN.0b013e3181d785d5. PMID 20431360
- [Derived] Palmas W, Shea S, Starren J, Teresi JA, Ganz ML, Burton TM, Pashos CL, Blustein J, Field L, Morin PC, Izquierdo RE, Silver S, Eimicke JP, Lantigua RA, Weinstock RS; IDEATel Consortium. Medicare payments, healthcare service use, and telemedicine implementation costs in a randomized trial comparing telemedicine case management with usual care in medically underserved participants with diabetes mellitus (IDEATel). J Am Med Inform Assoc. 2010 Mar-Apr;17(2):196-202. doi: 10.1136/jamia.2009.002592. PMID 20190064
- [Derived] Morin PC, Wolff LT, Eimicke JP, Teresi JA, Shea S, Weinstock RS. Record media used by primary care providers in medically underserved regions of upstate New York was not pivotal to clinical result in the Informatics for Diabetes Education and Telemedicine (IDEATel) project. Inform Prim Care. 2009;17(2):103-12. doi: 10.14236/jhi.v17i2.722. PMID 19807952
- [Derived] Sandberg J, Trief PM, Izquierdo R, Goland R, Morin PC, Palmas W, Larson CD, Strait JG, Shea S, Weinstock RS. A qualitative study of the experiences and satisfaction of direct telemedicine providers in diabetes case management. Telemed J E Health. 2009 Oct;15(8):742-50. doi: 10.1089/tmj.2009.0027. PMID 19780691
- [Derived] Shea S, Weinstock RS, Teresi JA, Palmas W, Starren J, Cimino JJ, Lai AM, Field L, Morin PC, Goland R, Izquierdo RE, Ebner S, Silver S, Petkova E, Kong J, Eimicke JP; IDEATel Consortium. A randomized trial comparing telemedicine case management with usual care in older, ethnically diverse, medically underserved patients with diabetes mellitus: 5 year results of the IDEATel study. J Am Med Inform Assoc. 2009 Jul-Aug;16(4):446-56. doi: 10.1197/jamia.M3157. Epub 2009 Apr 23. PMID 19390093
- [Derived] Shea S; IDEATel Consortium. The Informatics for Diabetes and Education Telemedicine (IDEATel) project. Trans Am Clin Climatol Assoc. 2007;118:289-304. PMID 18528511
- [Derived] Trief PM, Teresi JA, Izquierdo R, Morin PC, Goland R, Field L, Eimicke JP, Brittain R, Starren J, Shea S, Weinstock RS. Psychosocial outcomes of telemedicine case management for elderly patients with diabetes: the randomized IDEATel trial. Diabetes Care. 2007 May;30(5):1266-8. doi: 10.2337/dc06-2476. Epub 2007 Feb 26. No abstract available. PMID 17325261

RESULTS

PARTICIPANT FLOW:
Groups:
- Telemedicine Case Management: Telemedicine case management was performed through regular video-calls between a nurse case manager and the participant, with upload of blood glucose and blood pressure data (taken by the participant) through the telemedicine unit.
- Usual Care: Usual care consisted of continuing routine medical care, as prior to enrollment. Thus, diabetes management was performed by the participant's Primary Care Provider.
Period: Overall Study
Arm/Group | Telemedicine Case Management | Usual Care
Started | 844 | 821
Completed | 729 | 716
Not Completed | 115 | 105

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telemedicine Case Management | Usual Care | Total
Number analyzed (Participants) | 844 | 821 | 1665
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (6.5) | 70.9 (6.8) | 70.8 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 536 | 510 | 1046
  Male | 308 | 311 | 619

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c Levels
Time Frame: 5 years
Measure: Mean (Standard Error); unit: A1c percentage
Arm/Group | Telemedicine Case Management | Usual Care
Number analyzed (Participants) | 844 | 821
A1c percentage | 7.09 (0.06) | 7.38 (0.06)

2. Primary Outcome: Blood Pressure Levels
Time Frame: 5 years
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Telemedicine Case Management | Usual Care
Number analyzed (Participants) | 844 | 821
mmHg | 135.83 (0.87) | 140.15 (0.86)

3. Primary Outcome: Serum Lipids Levels; Low-density Lipoprotein (LDL)-Cholesterol
Time Frame: 5 years
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Telemedicine Case Management | Usual Care
Number analyzed (Participants) | 844 | 821
mg/dL | 91.13 (1.43) | 94.97 (1.40)

ADVERSE EVENTS:
Arm/Group | Telemedicine Case Management | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/844 | 0/821
Other Adverse Events (participants affected / at risk) | 0/844 | 0/821

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes